CLINICAL TRIAL: NCT01256632
Title: Evaluation of the Effect of Vitreous Composition Determined by Ultrasound and Optical Coherence Tomography (OCT) on Ranibizumab Therapy
Acronym: PVD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vision Research Foundation (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Michael T. Trese, M.D., DIrector of the Vision Research Foundation, Vision Research Foundation
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: FVF4316s
Record Dates: First submitted 2010-12-02; First posted 2010-12-08 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subfoveal CNV, secondary to AMD with PVD (Active Comparator): 20 eyes with Subfoveal Choroidal Neovascularization, secondary to Age Related Macular Degeneration, with Posterior Vitreous Detachment (PVD Positive). All study eyes will receive 0.5mg, of intravitreous monthly injections of Ranibizumab, for four initial doses,(Day 0, Month 1, Month 2, and Month 3),with scheduled follow-up visits monthly for 12 months. Re-treatment after.
  Interventions: Drug: Ranibizumab
- Subfoveal CNV, secondary to AMD w/o PVD (Active Comparator): 20 eyes with Subfoveal Choroidal Neovascularization, secondary to Age Related Macular Degeneration, without Posterior Vitreous Detachment (PVD Negative). All study eyes will receive 0.5mg, of intravitreous monthly injections of Ranibizumab, for four initial doses,(Day 0, Month 1, Month 2, and Month 3),with scheduled follow-up visits monthly for 12 months. Re-treatment after the first 4 injections, will be on an as needed basis, based on predefined criteria.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — All study eyes will receive 0.5mg, of intravitreous monthly injections of ranibizumab, for four initial doses,(Day 0, Month 1, Month 2, and Month 3),with scheduled follow-up visits monthly for 12 months. Re-treatment after.
  Other Names: Lucentis

SUMMARY:
The primary objective:

*To measure the difference in the number of Ranibizumab therapies needed in 12 months in the Posterior Vitreous Detachment (PVD) positive and Posterior Vitreous Detachment (PVD) negative group.

Secondary Objective:

* To measure the mean change in visual acuity from Baseline to Month 12.
* To measure the mean change in central retinal thickness per OCT from Baseline to Month 12

DETAILED DESCRIPTION:
This is an open-label study, of intravitreally administered Ranibizumab in eyes with Age-related Macular Degeneration (AMD), specifically looking at the correlation between the presence of Posterior Vitreous Detachment(PVD) and the number of intravitreal injections of Ranibizumab required. 40 subjects from the offices of Vision Research Foundation will be enrolled in this study. Subjects will be assigned to either a Posterior Vitreous Detachment (PVD) positive group or a Posterior Vitreous Detachment (PVD) negative group based on a pre-treatment ultrasound. A maximum of 20 subjects in each group will be enrolled. Subject accrual into the trial is expected to be completed within 6 months.

All study eyes will receive 0.5mg, of intravitreous monthly injections of Ranibizumab, for four initial doses,(Day 0, Month 1, Month 2, and Month 3),with scheduled follow-up visits monthly for 12 months. Re-treatment after the first 4 injections, will be on an as needed basis, based on predefined criteria. Eyes will be evaluated with a full ocular examination, visual acuity measurement (ETDRS chart at a distance of 4 meters),OCT,FA,Fundus Photos, B-scan Ultrasound and subject adverse event monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Subjects of either gender, Age greater than or equal to 50 years
* Best corrected visual acuity in the study eye between 20/25 and 20/320
* Subfoveal choroidal neovascularization, secondary to age related macular degeneration
* Total lesion size less than 4 disc diameters
* Any subretinal hemorrhage must comprise no more than 50% of total lesion size.
* Clear ocular media and adequate papillary dilation to permit good quality stereoscopic fundus photography
* Ability to return for all study visits

Exclusion Criteria:

* Pregnancy (positive pregnancy test)or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel,an IUD,or contraceptive hormone implant or patch.
* Patients with any form of prior eye treatment for AMD including: Photodynamic Therapy, anti-VEGF Therapy, Laser, Vitreoretinal surgery
* Had ocular surgery within the past 60 days in study eye
* Concurrent use of more than two therapies for glaucoma
* Uncontrolled glaucoma in the study eye(defined as intraocular pressure>30mm Hg despite treatment with anti-glaucoma medication)
* Concurrent use of systemic anti-VEGF agents
* Has active infection in the study eye(s)
* Inability to obtain photographs to document CNV
* Has received investigational therapy within 60 days prior to study entry
* Patients with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
* Has other conditions the investigator considers to be sound reasons for exclusion(e.g., lack of motivation, history of poor compliance, concomitant illnesses, personality disorder, mental condition, drug abuse, use of neuroleptics, physical or social condition predicting difficulty in long-term follow-up).
* Has an allergy to sodium fluorescein dye
* Inability to comply with study or follow-up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Difference in the number of Ranibizumab therapies needed in 12 months in the Posterior Vitreous Detachment positive and Posterior Vitreous Detachment negative group | 12 months

SECONDARY OUTCOMES:
Mean change in visual acuity from Baseline to Month 12 | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Trese, MD, Principal Investigator — Vision Research Foundation
Locations (1):
- Vision Research Foundation, Royal Oak, Michigan, United States